CLINICAL TRIAL: NCT02881814
Title: Evaluation of the Impact of Lung and Diaphragm Ultrasound Findings on Clinical Decisions for Chest Physiotherapy in Patients Hospitalized in Intensive Care Units
Brief Title: UltraSound for Accurate Decisions in Chest PhysioTherapy
Acronym: US-ADEPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Collaborators: Hopital Forcilles (Other); Centre Hospitalier Universitaire Dijon (Other); St Vincent's Hospital, Sydney (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: US-ADEPT
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Critical Illness; Respiratory Disease
Keywords: Lung ultrasound; Chest physiotherapy; Decision-making process; Diagnostic
MeSH Terms: conditions — Critical Illness; Respiration Disorders; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lung ultrasound and clinical decision (Experimental): Clinical assessment and choice of chest physiotherapy treatmetn performed by the clinical physiotherapist, followed by a comprehensive lung and diaphragm ultrasonography. After ultrasonography, the clinical physiotherapist is asked what CPT treatment he was going finally to implement, and explain the reasons for change, if any.
  Interventions: Diagnostic Test: Lung and diaphragm ultrasound
- Mechanically ventilated patients (Experimental): In case of mechanically ventilated patient at St. Vincent Hospital (Sydney, Australia), LUS scan will be performed immediately following intubation. Additionnal LUS scans will be performed 72h after intubation and Immediately prior to or following extubation.
  Interventions: Diagnostic Test: Lung and diaphragm ultrasound; Diagnostic Test: Lung and diaphragm ultrasound in MV patients

INTERVENTIONS:
Diagnostic Test: Lung and diaphragm ultrasound — The ultrasound physiotherapist/operator performs a lung and diaphragm ultrasound. He is blinded to the patient's status and clinical physiotherapist examination. He/she is not involved in patient management or patient clinical decision-making. The ultrasound findings are recorded in the LUS report. The LUS report is reported to the clinical physiotherapist and to the intensivist. The ultrasound diagnosis(es) is recorded.
Diagnostic Test: Lung and diaphragm ultrasound in MV patients — In case of mechanically ventilated patient at St. Vincent Hospital (Sydney, Australia), LUS scan will be performed immediately following intubation. Additionnal LUS scans will be performed 72h after intubation and Immediately prior to or following extubation.
  Arms: Mechanically ventilated patients

SUMMARY:
Introduction: Physiotherapist usually uses a clinical examination, including auscultation, an analysis of blood gasses and chest imaging to determine the indication for chest physiotherapy, to choose the treatment protocol and evaluate the efficacy of the management. Lung ultrasound (LUS) presents greater accuracy than chest X-ray in the diagnosis of lung deficiencies interesting the physiotherapist. So, it could allow the physiotherapist to determine the indication for chest physiotherapy and thus avoid unnecessary or inappropriate treatments. No study has evaluated the impact of LUS on clinical decisions in chest physiotherapy in ICU patients.

Objective: To evaluate the impact of using the results of lung and diaphragm US on clinical decisions in chest physiotherapy in hypoxemic patients hospitalized in ICU.

Method: The physiotherapist carries out a clinical examination and analyses the complementary tests (chest X-ray, chest CT-scan and blood gasses if available). Following the examination, he will put forward one or several hypotheses concerning the respiratory deficiency and will confirm or not the indication for chest physiotherapy. If respiratory physiotherapy is indicated, the physiotherapist will specify the protocol.

A lung and diaphragm US will be done following the evaluation of the clinical physiotherapist, and will make it possible to answer the question: are the results of the lung and diaphragm US compatible with the hypotheses put forward? The LUS report will be given to the clinical physiotherapist. He will specify the respiratory physiotherapy protocol according to the results of the US-scan.

The modification of the clinical decision will be assessed with the Net Reclassification Index (NRI).

Expected results: We expect that decisions for chest physiotherapy will be modified by LUS. The expected benefit for patients is therefore that they will be given a chest physiotherapy protocol that is better suited to the type of respiratory deficiency they are suffering from.

DETAILED DESCRIPTION:
Research hypothesis The lung and diaphragm ultrasound findings provided to the physiotherapist will modify his/her clinical decision-making in regards to chest physiotherapy treatment in the critical care patient.

Objectives Principal objective The principal objective of this study is to evaluate the impact of using the results of lung and diaphragm US on clinical decisions by physiotherapists regarding chest physiotherapy in patients hospitalized in an ICU.

Secondary objectives

1. Determine the accuracy of physiotherapist diagnosis of lung pathology using routine clinical assessment versus LUS findings;
2. Determine the frequency of change in chest physiotherapy treatment with the addition of LUS results to clinical assessment;
3. Determine the frequency of change in medical treatment (determined by intensivist) following the addition of LUS results to clinical assessment findings.
4. Evaluate the diagnostic accuracy of LUS in predicting duration of mechanical ventilation and mortality.

Methodology:

Type of study This is a multi-centre prospective (patients enrolled on admission) interventional study evaluating a routine assessment/treatment. The study intends to assess the impact of lung and diaphragm ultrasound on the usual physiotherapist's clinical decision-making process. Each included patient will be clinically assessed by a clinical physiotherapist, and then will have a lung and diaphragm ultrasound by another physiotherapist/operator blinded to the clinical assessment findings. The lung and diaphragm ultrasound findings will then be presented to both the intensivist and clinical physiotherapist to evaluate the impact on the independent clinical decision-making by both the intensivist and physiotherapist.

Data collections

The following data will be collected:

* Demographic: age, sex, BMI, smoking, alcohol consumption, history of cirrhosis, diabetes or a chronic respiratory disease, heart failure;
* Reason for hospitalization, medical diagnosis if different;
* Treatments: hypnotics, opiates, steroids and anti-hypertensives, oxygen therapy, mechanical ventilation, NIV, tracheotomy;
* Duration of mechanical ventilation
* Duration of ICU stay
* Vital signs: RR, HR, PA, SpO2, RASS, Glasgow;
* Clinical hypotheses of the clinical physiotherapist;
* LUS findings;
* Choice of chest physiotherapy protocol (before and after ultrasonography).

Nature of the routine care to be evaluated Procedure 1: Decision-making process in chest physiotherapy The clinical physiotherapist is the physiotherapist who manages patients in the CCU.

As soon as chest physiotherapy is prescribed, the physiotherapist carries out a clinical examination and analyses the complementary tests (chest X-ray, chest CT-scan and blood gasses if available). He/she also consults the patient's medical record to find out the reason for admission to the CCU and the medical diagnosis if the critical care physician has made one. Following the examination, he/she will put forward one or several hypotheses concerning the respiratory deficiency (and not the disease - medical diagnosis) and will confirm or not the indication for chest physiotherapy. If respiratory physiotherapy is indicated, the physiotherapist will specify the protocol.

A lung and diaphragm US will be done (see below) following the evaluation of the clinical physiotherapist, and will make it possible to answer the question: are the results of the lung and diaphragm US compatible with the hypotheses put forward? The LUS report will be given to the clinical physiotherapist. It will specify the respiratory physiotherapy protocol according to the results of the US-scan.

Procedure 2: lung and diaphragm US The LUS will be performed by the physiotherapist/operator, who will be blinded to the clinical evaluation of the clinical physiotherapist and the patient's status. The operator will not take part in the management of the patients concerned. The semiology of lung and diaphragm US is described. The following syndromes will be searched for: normal profile, alveolar-interstitial syndrome, pulmonary consolidation, pleural effusion, pneumothorax and diaphragm dysfunction. The physiotherapist/operator will write a detailed LUS-scan report, which will be given to the clinical physiotherapist. It will include the LUS diagnosis and describe the signs observed in the different regions of the chest. The clinical physiotherapist is trained to interpret LUS reports.

In case of mechanically ventilated patient at St. Vincent Hospital (Sydney, Australia), LUS scan will be performed immediately following intubation. Additionnal LUS scans will be performed 72h after intubation and Immediately prior to or following extubation.

Number of patients to recruit and duration of participation for each patient Given the high prevalence of hypoxemia in ICUs, the systematic respiratory assessment in these patients by the physiotherapist and our relatively non-restrictive inclusion criteria, we believe we can recruit more than 300 patients per year.

ELIGIBILITY:
Inclusion criteria

* Hypoxemia(SpO2/FiO2< 315 (15))(indication for chest physiotherapy)(cf. annexe 1);
* Medical prescription for chest physiotherapy;
* First session of chest physiotherapy;
* Chest X-ray<12h available;
* Physiotherapist/operator qualified in LUS available;
* Patient's consent.

Exclusion criteria

* Presence of a contra-indication for chest physiotherapy;
* Absence of hypoxemia;
* Absence of a prescription for chest physiotherapy;
* Absence of a chest X-ray < 12h from the time of physiotherapy assessment;
* Physiotherapist/operator qualified in LUS not available;
* Lung and diaphragm US not possible (surgical emphysema, dressing, scarring, drains etc.);
* Refusal of the patient or a relative to participate in the study;
* Patients to be discharged on the day of the study;
* Patients in palliative care;
* Withdrawal/limitations of medical care with impending death.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2024-04-14 (Estimated)

PRIMARY OUTCOMES:
Net Reclassification Index (NRI) | Hour 1
  Agreement (yes/no) between the lung and diaphragm US diagnosis and the clinical diagnosis and modification (yes/no) of the chest physiotherapy protocol

SECONDARY OUTCOMES:
Prediction of duration of mechanical ventilation | Final study visit
  Number of days with mechanical ventialtion
Prediction of mortality | Final study visit
  Vital status at the end of ICU hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Belaid Bouhemad, MD, PhD, Study Director — Centre Hospitalier Universitaire Dijon; Aymeric Le Neindre, PhD, Principal Investigator — Hopital Forcilles; George Ntoumenopoulos, PhD, Principal Investigator — St Vincent's Hospital
Locations (4):
- St Vincent's Hospital, Sydney, Australia
- France (3):
  - CHU de Dijon, Dijon
  - Hôpital Forcilles, Férolles-Attilly
  - Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be openly available in "figshare".
Supporting Information: SAP, Analytic Code
Time Frame: At publication.
Access Criteria: The data that support the findings of this study will be openly available

REFERENCES:
- [Result] Xirouchaki N, Georgopoulos D. Impact of lung ultrasound on clinical decision making in critically ill patients: response to O'Connor et al. Intensive Care Med. 2014 Jul;40(7):1063. doi: 10.1007/s00134-014-3316-6. Epub 2014 May 6. No abstract available. PMID 24797688
- [Result] Le Neindre A, Mongodi S, Philippart F, Bouhemad B. Thoracic ultrasound: Potential new tool for physiotherapists in respiratory management. A narrative review. J Crit Care. 2016 Feb;31(1):101-9. doi: 10.1016/j.jcrc.2015.10.014. Epub 2015 Oct 26. PMID 26613650
- [Result] Leech M, Bissett B, Kot M, Ntoumenopoulos G. Lung ultrasound for critical care physiotherapists: a narrative review. Physiother Res Int. 2015 Jun;20(2):69-76. doi: 10.1002/pri.1607. Epub 2014 Dec 29. PMID 25545613
- [Derived] Le Neindre A, Hansell L, Wormser J, Gomes Lopes A, Diaz Lopez C, Romanet C, Choukroun G, Nguyen M, Philippart F, Guinot PG, Buscher H, Bouhemad B, Ntoumenopoulos G. Thoracic ultrasound influences physiotherapist's clinical decision-making in respiratory management of critical care patients: a multicentre cohort study. Thorax. 2023 Feb;78(2):169-175. doi: 10.1136/thoraxjnl-2021-218217. Epub 2022 Mar 23. PMID 35321941

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-06-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT02881814/Prot_SAP_ICF_000.pdf